CLINICAL TRIAL: NCT01283919
Title: A Randomized, Two-treatment, Two-period, Two-sequence,Single Dose, Crossover Bioequivalence Study of Pantoprazole Sodium 40 mg Delayed Release Tablets (Dr. Reddy's Laboratories Ltd, India) to be Compared With Protonix® 40 mg (Pantoprazole Sodium) Delayed Release Tablets (Wyeth Laboratories, USA) in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Pantoprazole Sodium DR Tablets 40 mg of Dr. Reddy's Laboratories Limited Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice President-Research and Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PAN/23/87/04-05
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pantoprazole Sodium (Experimental): Pantoprazole Sodium DR Tablets 40 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Pantoprazole Sodium
- Protonix (Active Comparator): Protonix 40 mg DR Tablets of Wyeth Laboratories
  Interventions: Drug: Pantoprazole Sodium

INTERVENTIONS:
Drug: Pantoprazole Sodium — Pantoprazole Sodium DR Tablets 40 mg
  Other Names: Protonix DR Tablets 40 mg

SUMMARY:
To compare the single dose bioavailability of pantoprazole sodium 40 mg delayed release tablets (Dr. Reddy's Laboratories Ltd, India) with Protonix® 40 mg delayed release tablets (Wyeth Laboratories, USA) in 42 (+ 4 standby) healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
This is a Open label, balanced, randomized two-treatment, two-period,two-sequence, crossover bioequivalence study with at least 07 days washout period between each drug administration under fasting conditions.42 (+4 standby) healthy, adult, human subjects were enrolled. A single oral dose of40 mg of pantoprazole delayed release tablet will be administered along with 240 mL of drinking water after an overnight fast of at least 10 hours in each period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will provide written informed consent.
2. Subjects must be healthy human beings within 18-45 years of age (inclusive) weighing at least 50 kg.
3. Subjects must be within ±10% of ideal body weight in relation to height according to Life Insurance Corporation of India height-weight chart for non-medical cases.
4. Subjects must be of normal health as determined by medical history and physical examination performed within 15 days prior to the commencement of the study.
5. Have normal EcG, X-ray and vital signs.
6. Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
7. If subject is a female volunteer and

   1. Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
   2. is postmenopausal for at least 1 year.
   3. is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

1. Subjects incapable of understanding the informed consent.
2. Subjects with BP≤90/60 or BP≥140/90
3. History of hypersensitivity or idiosyncratic reaction to pantoprazole or other proton pump inhibitors.
4. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
5. Regular smoker who smokes more than ten cigarettes daily and has difficulty in abstaining from smoking for the duration of each study period.
6. Subjects who has taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within the past 30 days prior to start of clinical period.
7. History of any psychiatric illness, which may impair the ability to provide written, informed consent.
8. Subjects who have a history of alcohol or substance abuse within the last 5 years.
9. Subjects with clinically significant abnormal values of laboratory parameters.
10. Subjects who have participated in any other clinical investigation using experimental drug or had bled more than 350 mL in the past 3 months.
11. Subjects with positive urine screen for drugs of abuse.
12. Any subject in whom pantoprazole is contraindicated for medical reasons.
13. Female volunteers demonstrating a positive pregnancy screen.
14. Female volunteers who are currently breast-feeding.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Kulkarni, M.D, Principal Investigator — VimtaLabsLtd.
Locations (1):
- VimtaLabsLtd., Hyderabad, Andhrapradesh, India